The Effect of Preoperative Oral Carbohydrate Administration on Postoperative Glucometabolic Response, Subjective Well Being and Quality of Life in Patients **Undergoing Colorectal Surgery: A Randomized Controlled Double-Blind Study** 

Trial registration: NCT05402592

Date of the document: 06.03.2025

# Murat URKAN<sup>1</sup>, Cemile CELEBI<sup>2</sup>, Ulvi Mehmet MERAL<sup>3</sup>, Ikbal CAVDAR<sup>4</sup>

- <sup>1</sup> Associate Professor Doctor, Department of General Surgery, Acibadem Bodrum Hospital, Muğla, Turkey, murat.urkan@acibadem.com/ muraturkan@gmail.com ORCID: 0000-0002-3191-4724
- <sup>2</sup> Assistant Professor Doctor, PhD, Muğla Sıtkı Koçman University Faculty of Health Sciences, Department of Nursing, Department of Surgical Diseases Nursing, Muğla/Turkey, cemilecelebi@mu.edu.tr/ccelebi48@gmail.com ORCID:0000-0001-9960-7205
- <sup>3</sup> Doctor, Kayseri State Hospital, Department of General Surgery, Kayseri, Turkey, ulvimeral@yahoo.com ORCID: 0000-0001-7399-6353
- <sup>4</sup> Professor Doctor, Istanbul Atlas University, Faculty of Health Sciences, Department of Nursing, Istanbul, Turkey, ikbal.cavdar@atlas.edu.tr ORCID: 0000-0002-8242-6165
  - Corresponding author: Cemile ÇELEBİ/ cemilecelebi@mu.edu.tr /ccelebi48@gmail.com

## INTRODUCTION

Preoperative fasting has traditionally been a standard practice for patients undergoing elective surgery, primarily aimed at reducing the risk of pulmonary aspiration (1). However, prolonged fasting periods have been associated with increased preoperative anxiety, delayed surgical recovery, and heightened perioperative insulin resistance (PIR) (2,3). Surgical trauma, combined with prolonged fasting, exacerbates catabolic processes and triggers a metabolic stress response, leading to increased patient discomfort and complications (4,5). In response to these challenges, recent research and evidence-based guidelines have shifted focus toward minimizing the duration of preoperative fasting. Notably, the administration of oral carbohydrates in the preoperative period has been recommended to mitigate these adverse effects (6,7).

The Enhanced Recovery After Surgery (ERAS) protocols advocate for preoperative oral carbohydrate loading, particularly in patients undergoing elective colorectal surgery (6). Preoperative carbohydrate intake has been shown to modulate perioperative metabolism, reduce the stress response to surgical trauma, prevent complications, improve surgical outcomes, shorten hospital stays, and decrease postoperative morbidity and mortality (8–11). The International Society of Anaesthesia has confirmed the safety of oral carbohydrate intake, stating that it does not increase the risk of anesthesia-related complications. Furthermore, reducing the fasting period and administering carbohydrate-containing liquids have been shown to alleviate perioperative thirst, hunger, weakness, fatigue, anxiety, postoperative nausea and vomiting, and to promote intestinal peristalsis and shorter hospital stays (12–15). Despite these advancements, there remains a gap in the literature regarding the comprehensive impact of preoperative carbohydrate loading on postoperative quality of life and subjective well-being, particularly in the context of colorectal surgery. While previous studies have primarily focused on metabolic outcomes and clinical recovery parameters, the effects on

patient-reported outcomes such as quality of life and subjective well-being have not been thoroughly investigated. This study aims to address this gap by examining the effects of preoperative oral carbohydrate ingestion on postoperative glucometabolic response, subjective well-being, quality of life, and surgical clinical outcomes in patients undergoing colorectal surgery.

The originality of this study lies in its holistic approach to evaluating both clinical and patient-centered outcomes. By integrating traditional clinical metrics with patient-reported outcomes, this research provides a more comprehensive understanding of the benefits of preoperative carbohydrate loading. Furthermore, the study employs a double-blind, randomized controlled design, ensuring robust and unbiased results. The findings of this study have the potential to inform clinical practice by highlighting the multifaceted benefits of preoperative carbohydrate administration, thereby contributing to the optimization of perioperative care protocols.

# **Research Hypotheses**

- **H1-1:** Preoperative oral carbohydrate intake reduces postoperative insulin resistance in patients undergoing colorectal surgery.
- **H1-2:** Preoperative oral carbohydrate intake improves subjective well-being in patients undergoing colorectal surgery.
- **H1-3:** Preoperative oral carbohydrate intake enhances the quality of life in patients undergoing colorectal surgery.

### **METHODS**

## Participants and sampling

This prospective, randomized controlled double-blind study was conducted at the General Surgery Clinic of A University Hospital between January 2022 and April 2023. The sample size was determined based on an effect size calculation derived from a previous study by Yagci et al. (3), which reported a mean glucose level difference of 12.18 mg/dL between the

experimental and control groups. Using this data, the effect size (d) was calculated as 0.72. With a 95% confidence level (1-α) and 80% statistical power (1-β), the G\*Power software (version 3.1) was used to determine that a minimum of 25 participants per group (50 participants in total) would be required to detect significant differences between the groups.

The study population consisted of patients aged 18 years or older who were scheduled for elective colorectal surgery and had the capacity to provide informed consent. Participants were classified as American Society of Anesthesiologists (ASA) physical status I, II, or III. Exclusion criteria included patients diagnosed with diabetes, gastroesophageal reflux disease (GERD), severe liver or kidney failure, hiatal hernia, or those with oral nutrition difficulties. Additionally, emergency cases and patients classified as ASA IV or higher were excluded from the study.

# Randomization and blinding

Randomization was performed by a researcher who were not directly involved in the clinical aspects of the study, with a sequence generated by a computer program (<a href="https://www.random.org">https://www.random.org</a>) to assign 50 patients randomly to 2 groups in an unbiased manner. The list was kept secret from the patients and the researchers who registered and evaluated the patients until the final of the study. To maintain blinding, the study beverages were prepared in bottles of the same form by a nutrition company employee who was not actively engaged in the research process. Additionally, the statistical analysis was performed independently by an experienced statistician, who was not directly involved in the study.

## **Data collection**

The data were compiled via a personal interview with the participants, who were asked to complete a four-part evaluation form. This form was designed by the research team and based on the findings of relevant literature.

### **Observation indicators**

**Primary outcomes:** Reducing insulin resistance (below 2.5 mg/dl), shortening hospital stay, ensuring subjective well-being.

**Secondary outcomes:** The early return of bowel movements, shorter passing-gas time, and higher quality of life on the 30th day after surgery were observed in patients who received carbohydrate-rich drinks.

### **Interventions**

The study interventions were designed to evaluate the effects of preoperative carbohydrate intake on postoperative outcomes. Participants were divided into two groups: the intervention group (carbohydrate drink) and the control group (water). Both groups followed a standardized protocol, as outlined below:

**Intervention Group:** Patients in the intervention group were administered 800 mL of a carbohydrate-rich drink (12.5 g carbohydrate per 100 mL, containing 12% monosaccharides, 12% disaccharides, and 76% polysaccharides, with an osmolality of 285 mOsm/kg) until midnight on the day before surgery. Additionally, 400 mL of the same carbohydrate drink was given 2-3 hours before the surgical procedure (Figure 1).

**Control Group:** Patients in the control group received 800 mL of water until midnight on the day before surgery and 400 mL of water 2-3 hours before the procedure (Figure 1).

### **Data Collection:**

Data were collected in four main categories:

**Descriptive Characteristics:** Age, gender, education level, marital status, occupation, body mass index (BMI), smoking and alcohol use, presence of chronic diseases, ASA score, and clinical outcomes (time to first flatulence, first defecation, first oral feeding, first mobilization, and hospital stay).

**Laboratory Findings:** Gastric pH, gastric volume, and blood markers (glucose, insulin, cortisol, albumin, potassium, sodium, magnesium, and urea) were measured at specific time points (preoperatively and 24 hours postoperatively).

Subjective Well-Being: Postoperative comfort indicators (pain, thirst, hunger, dry mouth, nausea, vomiting, weakness, and anxiety) were assessed using a Visual Analog Scale (VAS). The VAS is a 10 cm horizontal or vertical line, with endpoints labeled "No Pain" (0) and "Unbearable Pain" (10). Patients mark their level of discomfort on the line, and the score is measured in centimeters. A score of 0 indicates no discomfort, 1-4 indicates mild discomfort, 5-6 indicates moderate discomfort, and 7-10 indicates severe discomfort (16). The VAS was administered at specific postoperative time points (e.g., 8, 12, and 24 hours) to evaluate changes in subjective well-being.

Quality of Life: The SF-36 Quality of Life Scale was used to evaluate eight health domains 30 days after surgery. The SF-36 is a self-reported questionnaire consisting of 36 items that assess physical functionality, social functionality, role limitations due to physical and emotional problems, mental health, vitality, pain, and general health perception. Each domain is scored from 0 to 100, with higher scores indicating better health-related quality of life (17). The SF-36 was administered 30 days postoperatively to assess the long-term impact of preoperative carbohydrate intake on patients' quality of life.

## **Application of the Intervention**

- Patients were informed about the study during their preoperative assessment and provided both verbal and written consent.
- Participants were instructed to maintain regular eating and sleeping patterns for three days prior to hospitalization.
- Blood samples were collected at four time points: before the morning dose, 40 minutes and 90 minutes after drink ingestion, and during anesthesia induction.

• Gastric residue was measured intraoperatively using a nasogastric or orogastric tube, and pH values were recorded using a urine pH meter.

## Statistical analysis

The statistical analysis was conducted via the IBM SPSS Statistics 26 software (IBM Corp., Armonk, NY, USA). The distribution of scores obtained from each continuous variable was investigated using a combination of descriptive, graphical and statistical methods. The Shapiro-Wilk test was employed to ascertain the normality of the scores obtained from a continuous variable utilising a statistical methodology. Categorical variable data are presented as frequencies (n, %), while continuous variable data are presented as means±standard deviations. In order to make comparisons between two groups in relation to normally distributed quantitative variables, an independent sample t-test was employed. Conversely, when the variables in question were not normally distributed, a Mann-Whitney U test was used. To compare qualitative data between groups, chi-square tests (including the Yates correction and Fisher's exact test) were employed. The results were evaluated for statistical significance within the 95% confidence interval, with p<0.05 deemed significant.

## **RESULTS**

# Patient descriptive characteristics

The mean age of the patients included in the study was 66.64±10.26 years, 52% were male, the average BMI level was 25.44±3.37, 84% were married, and 74% were primary education. It was determined that 30% of the participants smoked, 20% consumed alcohol and 72% had a chronic disease. No statistically significant differences were observed in the distribution of the descriptive characteristics of the patients according to the research groups (Table 1).

# **Postoperative features**

In the preoperative period, a comparison was made among the patients in the experimental group and those in the control group in the postoperative period; gas, stool passage, transition

to oral feeding, mobility, and length of stay were statistically significantly shorter (p<0.001) (Table 2).

## Laboratory findings

The plasma glucose level in the patients in the experimental group was found to be statistically significantly lower in the preoperative period (p=0.002). However, plasma glucose (p<0.001) and insulin (p = 0.029) levels were determined to be higher in the measurement made during anaesthesia induction. Preoperative CRP (p=0.013) and both preoperative and postoperative 24th hour urea (p=0.034 and p=0.040) levels were significantly lower in the patients in the experimental group; It was determined that preoperative magnesium (p=0.025), postoperative 24th hour potassium (p=0.035) and both preoperative and postoperative 24th hour albumin (p=0.003 and p<0.001) levels were significantly higher (Table 2).

# Life quality

When the SF-36 quality of life scale scores of the patients were examined, except for the vitality and emotional role difficulty sub-dimensions (p>0.05), all other sub-dimensions were different between the research groups (p<0.01 and p<0.001). It was demonstrated that the quality of life, as measured by physical functionality, physical role difficulties, general health, pain, social function and mental health, was significantly superior in the patients in the experimental group. (Table 2).

## Patients' subjective well-being-related characteristics

Thirst at the 8th postoperative hour (p=0.018); The level of hunger (p=0.005) at the 12th hour and pain (p=0.007) at the 24th hour in the patients in the experimental group; It was established that the level of fatigue at the 12th and 24th postoperative hours (p<0.001) was significantly better only in the in the control group patients (Table 3).

# Ethics approval and consent to participate

The single-center, randomized controlled double-blind study was registered in the ClinicalTrials database (https://clinicaltrials.gov, NCT05402592). Prior to the commencement of the research, approval was sought and obtained from the Mugla Sitki Kocman University Clinical Research Ethics Committee (22.12.2021-27/II) and the chief physician of the hospital where the research would be conducted. In conducting the research, the authors adhered to the principles set forth in the Declaration of Helsinki. Written and verbal informed consent was obtained from all patients participating in the study. It was explained to the patients that all data would be confidential and that they had the right to withdraw from the study at any time. This research was conducted in accordance with Consolidated Standards of Reporting Trials (CONSORT) 2010 guidelines.

Table 1: Patient descriptive characteristics

Total Experiment

| (n=50) | (n=25) | (n=25) | Test value | <i>P</i> -value |
|---|---|---|---|---|
| 66.64±10.26 | 67.04±7.63 | 66.24±12.51 | 0.273ª | 0.786 |
| $25.44 \pm 3.37$ | $25.86 \pm 3.81$ | $25.02\pm2.89$ | $0.886^{\mathrm{a}}$ | 0.380 |
| | | | $0.721^{b}$ | 0.396 |
| 24(48.0) | 14(56.0) | 10(40.0) | | |
| 26(52.0) | 11(44.0) | 15(60.0) | | |
| | | | _c | 0.999 |
| 42(84.0) | 21(84.0) | 21(84.0) | | |
| 8(16.0) | 4(16.0) | 4(16.0) | | |
| | | | $0.884^{c}$ | 0.804 |
| 37(74.0) | 18(72.0) | 19(76.0) | | |
| 6(12.0) | 4(16.0) | 2(8.0) | | |
| 7(14.0) | 3(12.0) | 4(16.0) | | |
| | | | $0.000^{b}$ | 0.999 |
| 15(30.0) | 7(28.0) | 8(32.0) | | |
| 35(70.0) | 18(72.0) | 17(68.0) | | |
| | | | _c | 0.289 |
| 10(20.0) | 7(28.0) | 3(12.0) | | |
| 40(80.0) | 18(72.0) | 22(88.0) | | |
| | | | $2.480^{b}$ | 0.115 |
| 36(72.0) | 15(60.0) | 21(84.0) | | |
| | 25.44±3.37<br>24(48.0)<br>26(52.0)<br>42(84.0)<br>8(16.0)<br>37(74.0)<br>6(12.0)<br>7(14.0)<br>15(30.0)<br>35(70.0)<br>10(20.0)<br>40(80.0) | 66.64±10.26 67.04±7.63<br>25.44±3.37 25.86±3.81<br>24(48.0) 14(56.0)<br>26(52.0) 11(44.0)<br>42(84.0) 21(84.0)<br>8(16.0) 4(16.0)<br>37(74.0) 18(72.0)<br>6(12.0) 4(16.0)<br>7(14.0) 3(12.0)<br>15(30.0) 7(28.0)<br>35(70.0) 18(72.0)<br>10(20.0) 7(28.0)<br>40(80.0) 18(72.0) | 66.64±10.26 67.04±7.63 66.24±12.51 25.44±3.37 25.86±3.81 25.02±2.89 24(48.0) 14(56.0) 10(40.0) 26(52.0) 11(44.0) 15(60.0) 42(84.0) 21(84.0) 21(84.0) 8(16.0) 4(16.0) 4(16.0) 37(74.0) 18(72.0) 19(76.0) 6(12.0) 4(16.0) 2(8.0) 7(14.0) 3(12.0) 4(16.0) 15(30.0) 7(28.0) 8(32.0) 35(70.0) 18(72.0) 17(68.0) 10(20.0) 7(28.0) 3(12.0) 40(80.0) 18(72.0) 22(88.0) | 66.64±10.26 67.04±7.63 66.24±12.51 0.273° 25.44±3.37 25.86±3.81 25.02±2.89 0.886° 0.721° 24(48.0) 14(56.0) 10(40.0) 26(52.0) 11(44.0) 15(60.0) 42(84.0) 21(84.0) 21(84.0) 8(16.0) 4(16.0) 4(16.0) 6(12.0) 4(16.0) 2(8.0) 7(14.0) 3(12.0) 4(16.0) 15(30.0) 7(28.0) 8(32.0) 35(70.0) 18(72.0) 17(68.0) -c 10(20.0) 7(28.0) 3(12.0) 40(80.0) 18(72.0) 22(88.0) 2.480° |

p>0.05, a: Independent samples t test, b: Chi-square test with Yates correction, c: Fisher's exact testi, SD:Standard deviation

Table 2: Some laboratory, quality of life and other postoperative findings of the patients

| | | Experiment | Control | | |
|---|---|---|---|---|---|
| | <b>Total (n=50)</b> | (n=25) | (n=25) | | |
| Variables | Mean±SD | Mean±SD | Mean±SD | Test value | <i>P</i> -value |
| Gas output | 43.30±5.12 | 40.60±4.52 | 46.00±4.22 | -4.010a | <0.001* |
| Stool output | $75.24 \pm 10.71$ | $68.64 \pm 7.94$ | $81.84 \pm 8.97$ | -4.721 <sup>a</sup> | <0.001* |
| Oral nutrition | $46.12 \pm 4.93$ | 43.80±4.84 | 48.44±3.87 | -3.675a | <0.001* |
| Mobilisation | $12.58 \pm 1.64$ | 12.16±1.77 | 13.00±1.41 | 1.853 <sup>b</sup> | 0.070 |
| <b>Duration of postoperative</b> | | | | | |
| hospitalisation | $12.48 \pm 3.36$ | 10.64±1.52 | 14.32±3.69 | -4.494 <sup>a</sup> | <0.001* |
| <b>HOMA-IR score</b> | $1.83 \pm 0.52$ | $1.70 \pm 0.41$ | $1.97 \pm 0.59$ | -1.951a | 0.051 |
| Gastric pH | 4.76±5.72 | 5.59±8.04 | 3.94±0.92 | -0.223ª | 0.823 |
| Gastric volume | $0.37 \pm 0.06$ | $0.37 \pm 0.05$ | $0.37 \pm 0.07$ | 0.211 <sup>b</sup> | 0.834 |
| Plasma-glucose | | | | | |
| Preoperative | 87.50±16.30 | 80.24±7.66 | 94.75±19.35 | -3.150a | 0.002* |
| 40.min | $95.86 \pm 17.70$ | 91.04±10.67 | 100.67±21.84 | -1.400a | 0.162 |
| 90.min | $103.04\pm20.83$ | 105.04±21.02 | 101.04±20.87 | -1.399a | 0.162 |
| Anaesthesia induction | 115.63±22.26 | 123.80±18.96 | 107.47±22.66 | -3.611a | <0.001* |
| Plasma-insulin | | | | | |
| Preoperative | $8.54 \pm 1.69$ | $8.68\pm2.10$ | $8.40 \pm 1.19$ | -0.160a | 0.873 |
| 40.min | $9.18\pm2.40$ | $9.98\pm2.91$ | $8.37 \pm 1.40$ | -1.792a | 0.073 |
| 90.min | $10.64 \pm 4.79$ | 12.13±6.33 | $9.16\pm1.47$ | -1.679ª | 0.093 |
| Anaesthesia induction | $10.72 \pm 3.27$ | 11.91±4.16 | 9.68±1.71 | -2.184a | 0.029* |
| Plasma-cortisol | | | | | |
| Preoperative | $12.35 \pm 1.77$ | 12.08±2.17 | 12.60±1.29 | 1.024 <sup>b</sup> | 0.311 |
| 40.min | 14.27±4.95 | 15.25±6.85 | 13.32±1.46 | -0.071 <sup>a</sup> | 0.943 |
| 90.min | 14.94±4.91 | $15.67 \pm 6.78$ | 14.24±1.79 | $-0.789^{a}$ | 0.430 |
| Anaesthesia induction | 15.13±2.56 | 15.32±3.51 | 14.96±1.23 | -1.008 <sup>a</sup> | 0.313 |
| CRP | | | | | |

| Preoperative | 29.76±72.18 | 4.61±11.61 | 54.91±95.83 | -2.484a | 0.013* |
|---|---|---|---|---|---|
| Postoperative 24th hour | 95.96±81.83 | 73.33±48.74 | 118.58±101.14 | -1.106a | 0.269 |
| Albumin | | | | | |
| Preoperative | 40.61±7.16 | 43.64±3.28 | 37.57±8.64 | -2.935a | 0.003* |
| Postoperative 24th hour | 36.89±7.54 | 40.72±4.13 | 33.07±8.28 | 4.135 <sup>b</sup> | <0.001* |
| Potassium | | | | | |
| Preoperative | 4.30±0.48 | 4.32±0.47 | 4.29±0.49 | 0.262 <sup>b</sup> | 0.795 |
| Postoperative 24th hour | 4.19±0.46 | 4.35±0.36 | 4.04±0.51 | -2.110 <sup>a</sup> | 0.035* |
| Sodium | | | | | |
| Preoperative | 139.73±2.49 | 139.80±2.33 | 139.65±2.68 | 0.211 <sup>b</sup> | 0.834 |
| Postoperative 24th hour | 140.34±2.26 | 140.20±1.44 | 140.48±2.89 | 0.434 <sup>b</sup> | 0.667 |
| Magnesium | | | | | |
| Preoperative | 2.26±0.54 | 2.47±0.62 | $2.05 \pm 0.36$ | -2.244a | 0.025* |
| Postoperative 24th hour | 2.20±0.53 | $2.34 \pm 0.58$ | $2.05\pm0.44$ | -1.569ª | 0.117 |
| Urea | | | | | |
| Preoperative | 26.33±12.17 | 23.01±5.65 | 29.65±15.74 | -2.125 <sup>a</sup> | 0.034* |
| Postoperative 24th hour | 26.74±25.68 | 20.84±4.72 | 32.64±35.38 | -2.057ª | 0.040* |
| SF-36 | | | | | |
| Physical functioning | $71.70 \pm 17.46$ | 82.00±11.81 | $61.40 \pm 16.17$ | -4.357 <sup>a</sup> | <0.001* |
| Role limitations due to | | | | | |
| physical health | 50.00±33.12 | $63.00 \pm 30.72$ | $37.00 \pm 30.72$ | -2.770 <sup>a</sup> | 0.006* |
| Pain | 67.75±13.18 | $73.20 \pm 13.95$ | $62.30\pm9.92$ | -3.467ª | 0.001* |
| General health | $61.40 \pm 14.81$ | $68.80 \pm 15.09$ | $54.00 \pm 10.31$ | -4.171 <sup>a</sup> | <0.001* |
| Vitality | $69.40 \pm 12.23$ | 72.20±13.77 | $66.60\pm9.97$ | -1.637 <sup>a</sup> | 0.102 |
| Social functioning | $60.25 \pm 21.23$ | 71.00±22.16 | $49.50 \pm 13.73$ | -3.791ª | <0.001* |
| Role limitations due to | | | | | |
| emotional health | $80.00\pm29.35$ | 81.33±27.35 | 78.67±31.74 | -0.133ª | 0.894 |
| Mental health | $78.48 \pm 10.28$ | 83.36±7.36 | 73.60±10.58 | -3.336ª | 0.001* |

<sup>\*</sup>p<0.05, a=Mann-Whitney U Test, b=Independent Samples Test, SD=Standard deviation

Table 3: Subjective well-being-related characteristics of patients

| | | A + 0 < 00 a | related characterist | Postop 8th | Postop 12th | Postop 24th |
|---|---|---|---|---|---|---|
| | | At 06.00 a.m. | Preop | hour | hour | hour |
| Variables | Grup | Mean±SD | Mean±SD | Mean±SD | Mean±SD | <b>Mean±SD</b> |
| Pain | Experiment | 0.16±0.55 | 0.12±0.44 | 1.80±1.41 | 3.24±0.72 | 3.12±0.97 |
| | Control | $0.00 \pm 0.00$ | $0.00 \pm 0.00$ | 1.44±1.42 | $3.24 \pm 0.97$ | $3.88 \pm 0.93$ |
| | Test value <sup>a</sup> | -1.429 | -1.429 | -0.915 | -0.023 | -2.675 |
| | <i>P</i> -value | 0.153 | 0.153 | 0.360 | 0.982 | 0.007* |
| Dehydration | Experiment | 0.24±0.66 | 0.12±0.44 | 1.00±1.91 | 2.92±1.50 | 4.76±1.05 |
| | Control | $0.00 \pm 0.00$ | $0.16 \pm 0.37$ | $1.52\pm1.23$ | $2.80 \pm 1.12$ | 4.32±1.52 |
| | Test value <sup>a</sup> | -2.063 | -0.792 | -2.360 | -0.627 | -0.529 |
| | <i>P</i> -value | 0.039* | 0.428 | 0.018* | 0.531 | 0.597 |
| Hunger | Experiment | 0.24±1.20 | 0.28±1.21 | 0.48±1.64 | 1.36±1.66 | 4.00±1.55 |
| | Control | $0.08 \pm 0.40$ | $0.52 \pm 0.71$ | $0.88 \pm 1.42$ | 2.52±1.76 | 4.08±1.38 |
| | Test value <sup>a</sup> | -0.029 | -2.509 | -1.830 | -2.802 | -0.409 |
| | <i>P</i> -value | 0.977 | 0.012* | 0.067 | 0.005* | 0.683 |
| Dry Mouth | Experiment | 0.20±0.50 | 0.16±0.62 | 1.92±1.50 | 3.44±1.19 | 5.08±1.08 |
| | Control | $0.00 \pm 0.00$ | $0.12 \pm 0.33$ | $2.24 \pm 1.09$ | $3.60\pm1.04$ | 4.88±1.67 |
| | Test value <sup>a</sup> | -2.063 | -0.410 | -1.779 | -1.322 | -0.454 |
| | <i>P</i> -value | 0.039* | 0.682 | 0.075 | 0.186 | 0.650 |
| Nausea | Experiment | 0.04±0.20 | 0.08±0.28 | $0.68\pm0.80$ | 1.44±0.96 | 1.96±1.27 |
| | Control | $0.04 \pm 0.20$ | $0.56 \pm 0.92$ | $1.08 \pm 1.08$ | $1.88 \pm 1.17$ | 2.16±1.37 |
| | Test value <sup>a</sup> | 0.000 | -2.225 | -1.276 | -1.552 | -0.627 |
| | <i>P</i> -value | 1.000 | 0.026* | 0.202 | 0.121 | 0.531 |
| Fatigue | Experiment | $0.00\pm0.00$ | $0.00\pm0.00$ | 1.56±1.19 | 2.76±0.97 | 3.84±1.25 |
| | Control | $0.00 \pm 0.00$ | $0.00 \pm 0.00$ | $1.12\pm1.09$ | $1.32\pm1.31$ | $1.72\pm1.54$ |
| | Test value <sup>a</sup> | 0.000 | 0.000 | -1.298 | -3.805 | -4.699 |
| | <i>P</i> -value | 1.000 | 1.000 | 0.194 | <0.001* | <0.001* |
| Anxiety | Experiment | 2.36±2.12 | 3.64±2.18 | 2.68±1.49 | 2.76±1.59 | 3.32±1.55 |
| | Control | 1.28±2.64 | 1.52±2.57 | 1.44±1.78 | $1.08\pm1.32$ | 1.04±1.59 |
| | Test value <sup>a</sup> | -2.425 | -3.153 | -2.560 | -3.569 | -4.278 |
| | <i>P</i> -value | 0.015* | 0.002* | 0.010* | <0.001* | <0.001* |

<sup>\*</sup>p<0.05, a=Mann-Whitney U Test, SD=Standard deviation



Figure 1: CONSORT Flow Diagram

## REFERENCES

- 1. Fawcett WJ, Thomas M. Pre-operative fasting in adults and children: clinical practice and guidelines. Anaesthesia [Internet]. 2019 Jan 30;74(1):83–8. Available from: https://associationofanaesthetists-publications.onlinelibrary.wiley.com/doi/10.1111/anae.14500
- 2. Pimenta GP, Aguilar-Nascimento JE de. Prolonged preoperative fasting in elective surgical patients: why should we reduce it? Nutr Clin Pr. 2014;29(1):22–8.
- 3. Yagci G, Can MF, Ozturk E, Dag B, Ozgurtas T, Cosar A, et al. Effects of preoperative carbohydrate loading on glucose metabolism and gastric contents in patients undergoing moderate surgery: a randomized, controlled trial. Nutr . 2008;24(3):212–6.
- 4. Akbarzadeh M, Eftekhari M, Shafa M, Alipour S, Hassanzadeh J. Effects of a new metabolic conditioning supplement on perioperative metabolic stress and clinical outcomes: a randomized, placebo-controlled trial. Iran Red Crescent Med J. 2016;18(1).
- Xu D, Zhu X, Xu Y, Zhang L. Shortened preoperative fasting for prevention of complications associated with laparoscopic cholecystectomy: a meta-analysis. J Int Med Res [Internet]. 2017;45(1):22–37. Available from: https://doi.org/10.1177/0300060516676411
- 6. Gustafsson UO, Scott MJ, Hubner M, Nygren J, Demartines N, Francis N, et al. Guidelines for Perioperative Care in Elective Colorectal Surgery: Enhanced Recovery After Surgery (ERAS®) Society Recommendations: 2018. Vol. 43, World Journal of Surgery. Springer New York LLC; 2019. p. 659–95.
- 7. Joshi GP, Abdelmalak BB, Weigel WA, Harbell MW, Kuo CI, Soriano SG, et al. 2023 American Society of Anesthesiologists Practice Guidelines for Preoperative Fasting:

- Carbohydrate-containing Clear Liquids with or without Protein, Chewing Gum, and Pediatric Fasting Duration—A Modular Update of the 2017 American Society of Anesthesio. Anesthesiology [Internet]. 2023 Feb 1;138(2):132–51. Available from: https://pubs.asahq.org/anesthesiology/article/138/2/132/137508/2023-American-Society-of-Anesthesiologists
- 8. Çilingir D, Candaş B. Cerrahi sonrası hızlandırılmış iyileşme protokolü ve hemşirenin rolü. J Anatolia Nurs Heal Sci. 2017;20(2):137–43.
- 9. Gümüs K, Pirhan Y, Aydın G, Keloglan S, Tasova V, Kahveci M. The Effect of Preoperative Oral Intake of Liquid Carbohydrate on Postoperative Stress Parameters in Patients Undergoing Laparoscopic Cholecystectomy: An Experimental Study. J PeriAnesthesia Nurs [Internet]. 2021 Oct;36(5):526–31. Available from: https://linkinghub.elsevier.com/retrieve/pii/S1089947220303701
- Hübner M, Addor V, Slieker J, Griesser A-C, Lécureux E, Blanc C, et al. The impact of an enhanced recovery pathway on nursing workload: A retrospective cohort study. Int J Surg. 2015;24(ptA):45–50.
- Pogatschnik C, Steiger E. Review of Preoperative Carbohydrate Loading. Nutr Clin Pr.
   2015 Oct 8;30(5):660–4.
- 12. Helminen H, Branders H, Ohtonen P, Saarnio J. Effect of pre-operative oral carbohydrate loading on recovery after day-case cholecystectomy. Eur J Anaesthesiol [Internet]. 2019 Aug;36(8):605–11. Available from: https://journals.lww.com/00003643-201908000-00008
- 13. Onalan E, Andsoy II, Ersoy OF. The Effect of Preoperative Oral Carbohydrate Administration on Insulin Resistance and Comfort Level in Patients Undergoing Surgery. J PeriAnesthesia Nurs [Internet]. 2019 Jun;34(3):539–50. Available from: https://linkinghub.elsevier.com/retrieve/pii/S1089947218302995

- 14. Pędziwiatr M, Pisarska M, Wierdak M, Major P, Rubinkiewicz M, Kisielewski M, et al. The Use of the Enhanced Recovery After Surgery (ERAS) Protocol in Patients Undergoing Laparoscopic Surgery for Colorectal Cancer A Comparative Analysis of Patients Aged above 80 and below 55. Polish J Surg [Internet]. 2015 Jan 1;87(11). Available from: https://www.degruyter.com/view/j/pjs.2015.87.issue-11/pjs-2016-0004/pjs-2016-0004.xml
- 15. Zhang Y, Min J. Preoperative Carbohydrate Loading in Gynecological Patients Undergoing Combined Spinal and Epidural Anesthesia. J Investig Surg [Internet]. 2020 Aug 8;33(7):587–95. Available from: https://www.tandfonline.com/doi/full/10.1080/08941939.2018.1546352
- 16. Yeşilyurt M, Faydalı S. AĞRI DEĞERLENDİRMESİNDE TEK BOYUTLU ÖLÇEKLERİN KULLANIMI. J Anatolia Nurs Heal Sci [Internet]. 2020 Sep 16; Available from: https://nursing-ataunipress.org/en/use-of-one-dimensional-scales-in-pain-assessment-13825
- 17. Koçyiğit H, Aydemir Ö, Ölmez N. Kısa Form36 (KF36)'nın Türkçe versiyonunun güvenilirliği ve geçerliliği. İlaç ve Tedavi Derg. 1999;12:102–6.
- 18. Lambert E, Carey S. Practice Guideline Recommendations on Perioperative Fasting. J Parenter Enter Nutr [Internet]. 2016 Nov 9;40(8):1158–65. Available from: https://aspenjournals.onlinelibrary.wiley.com/doi/10.1177/0148607114567713
- 19. Doo AR, Hwang H, Ki M-J, Lee J-R, Kim D-C. Effects of preoperative oral carbohydrate administration on patient well-being and satisfaction in thyroid surgery. Korean J Anesthesiol [Internet]. 2018 Oct 1;71(5):394–400. Available from: http://ekja.org/journal/view.php?doi=10.4097/kja.d.18.27143
- 20. Rizvanović N, Nesek Adam V, Čaušević S, Dervišević S, Delibegović S. A randomised controlled study of preoperative oral carbohydrate loading versus fasting in patients

- undergoing colorectal surgery. Int J Colorectal Dis. 2019 Sep 1;34(9):1551-61.
- 21. Nygren J, Thacker J, Carli F, Fearon KCH, Norderval S, Lobo DN, et al. Guidelines for Perioperative Care in Elective Rectal/Pelvic Surgery: Enhanced Recovery After Surgery (ERAS ® ) Society Recommendations. World J Surg [Internet]. 2013 Feb 6;37(2):285–305. Available from: https://onlinelibrary.wiley.com/doi/10.1007/s00268-012-1787-6
- 22. Lidder P, Thomas S, Fleming S, Hosie K, Shaw S, Lewis S. A randomized placebo controlled trial of preoperative carbohydrate drinks and early postoperative nutritional supplement drinks in colorectal surgery. Color Dis [Internet]. 2013 Jun 24;15(6):737–45. Available from: https://onlinelibrary.wiley.com/doi/10.1111/codi.12130
- 23. Şavluk ÖF, Kuşçu MA, Güzelmeriç F, Gürcü ME, Erkılınç A, Çevirme D, et al. Do preoperative oral carbohydrates improve postoperative outcomesin patients undergoing coronary artery bypass grafts? Turkish J Med Sci [Internet]. 2017;47:1681–6. Available from: https://journals.tubitak.gov.tr/medical/vol47/iss6/2
- 24. Pexe-Machado PA, de Oliveira BD, Dock-Nascimento DB, de Aguilar-Nascimento JE. Shrinking preoperative fast time with maltodextrin and protein hydrolysate in gastrointestinal resections due to cancer. Nutrition [Internet]. 2013 Jul;29(7–8):1054–9. Available from: https://linkinghub.elsevier.com/retrieve/pii/S0899900713000956
- 25. Yılmaz H, Gülen G, Atalan G, Taş C, Özbek Ö, Aytaç Ş, et al. The effects on surgery stress of preoperative oral carbohydrate intake of knee and hip replacement surgery. Anatol J Clin Investig. 2013;7(3):158–63.
- Yildiz H, Gunal SE, Yilmaz G, Yucel S. Oral Carbohydrate Supplementation Reduces
   Preoperative Discomfort in Laparoscopic Cholecystectomy. J Investig Surg [Internet].
   Apr 10;26(2):89–95. Available from:
   https://www.tandfonline.com/doi/full/10.3109/08941939.2012.699998

- Yi HC, Ibrahim Z, Abu Zaid Z, Mat Daud Z 'Azuan, Md. Yusop NB, Omar J, et al. Impact of Enhanced Recovery after Surgery with Preoperative Whey Protein-Infused Carbohydrate Loading and Postoperative Early Oral Feeding among Surgical Gynecologic Cancer Patients: An Open-Labelled Randomized Controlled Trial. Nutrients [Internet]. 2020 Jan 20;12(1):264. Available from: https://www.mdpi.com/2072-6643/12/1/264
- 28. Hamamoto H, Yamamoto M, Masubuchi S, Ishii M, Osumi W, Tanaka K, et al. The impact of preoperative carbohydrate loading on intraoperative body temperature: a randomized controlled clinical trial. Surg Endosc. 2018 Nov 1;32(11):4393–401.
- 29. Webster J, Osborne SR, Gill R, Chow CFK, Wallin S, Jones L, et al. Does Preoperative Oral Carbohydrate Reduce Hospital Stayα A Randomized Trial. AORN J. 2014 Feb;99(2):233–42.
- 30. Chaudhary NK, Sunuwar DR, Sharma R, Karki M, Timilsena MN, Gurung A, et al.

  The effect of pre-operative carbohydrate loading in femur fracture: a randomized controlled trial. BMC Musculoskelet Disord [Internet]. 2022 Aug 30;23(1):819.

  Available from:

  https://bmcmusculoskeletdisord.biomedcentral.com/articles/10.1186/s12891-022-05766-z
- 31. Cho E-A, Lee NH, Ahn J-H, Choi W-J, Byun J-H, Song T. Preoperative Oral Carbohydrate Loading in Laparoscopic Gynecologic Surgery: A Randomized Controlled Trial. J Minim Invasive Gynecol [Internet]. 2021 May;28(5):1086-1094.e1. Available from: https://linkinghub.elsevier.com/retrieve/pii/S1553465020311699
- 32. Singh BN, Dahiya D, Bagaria D, Saini V, Kaman L, Kaje V, et al. Effects of preoperative carbohydrates drinks on immediate postoperative outcome after day care laparoscopic cholecystectomy. Surg Endosc [Internet]. 2015 Nov 22;29(11):3267–72.

Available from: http://link.springer.com/10.1007/s00464-015-4071-7